CLINICAL TRIAL: NCT00000508
Title: Stanford Coronary Risk Intervention Project (SCRIP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 27; R01HL028292 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 1993-03

CONDITIONS: Cardiovascular Diseases; Coronary Arteriosclerosis; Coronary Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Diet, Reducing; Exercise; Diet, Fat-Restricted

INTERVENTIONS:
Behavioral: smoking cessation
Behavioral: diet, reducing
Behavioral: exercise
Behavioral: diet, fat-restricted

SUMMARY:
To determine whether modification of risk factors altered the rate of progression of coronary artery disease in arteries with mild atherosclerosis and no mechanical intervention in patients who had coronary bypass surgery or percutaneous transluminal coronary angioplasty (PTCA).

DETAILED DESCRIPTION:
BACKGROUND:

Because of difficulties with quantitative measurement and with feasibility of follow-up, few controlled studies prior to SCRIP had been completed to determine the impact of risk factor modification directly on the progression of coronary atherosclerosis in humans. Suggestive evidence existed from animal studies, especially in primates, that diet and exercise altered atherosclerosis as a result of risk modification. But these animal models did not accurately represent the potential for modifying the coronary atherosclerotic process in humans. Some indirect evidence had been developed in humans by studying arteries more accessible than the coronaries. In the several preliminary studies reported using coronary arteriography to study the impact of risk modification on atherosclerosis, the results had been encouraging but far from definitive. One angiographic follow-up study of vein bypass grafts and severely atherosclerotic coronary arteries reported improvement with lipid lowering therapy. None of these studies had included randomization of patients to systematic, intense, long-term risk reduction versus usual care with prospectively identified coronary artery segments with mild disease.

DESIGN NARRATIVE:

Randomized, fixed-sample. A total of 300 patients were randomized, 155 to usual care (UC) in the community and 145 to special intervention (SI). The SI group received intensive efforts directed at reducing or eliminating risk factors, including lowering LDL-cholesterol and increasing HDL-cholesterol, reducing blood pressure, eliminating cigarette smoking and obesity, increasing exercise, and decreasing stressful life experience. The major endpoint was the rate of coronary artery disease progression as measured by angiography, at baseline and at forty-eight months. Follow-up was for four years.

ELIGIBILITY:
Men and women, up to 75 years of age. Patients with coronary artery disease but no mechanical intervention on all major vessels.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1983-09; Study Completion 1993-03

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Alderman — Stanford University; Ronald Krauss — University of California

REFERENCES:
- [Background] Leung WH, Demopulos PA, Alderman EL, Sanders W, Stadius ML. Evaluation of catheters and metallic catheter markers as calibration standard for measurement of coronary dimension. Cathet Cardiovasc Diagn. 1990 Nov;21(3):148-53. doi: 10.1002/ccd.1810210305. PMID 2225049
- [Background] Burge C, Sanders W, Alderman EL. Anatomic and machine projection angles of various radiographic imaging systems used for cardiac angiography. Cathet Cardiovasc Diagn. 1991 Jan;22(1):64-74. doi: 10.1002/ccd.1810220116. PMID 1995179
- [Background] Maron DJ, Fair JM, Haskell WL. Saturated fat intake and insulin resistance in men with coronary artery disease. The Stanford Coronary Risk Intervention Project Investigators and Staff. Circulation. 1991 Nov;84(5):2020-7. doi: 10.1161/01.cir.84.5.2020. PMID 1934376
- [Background] Haskell WL, Alderman EL, Fair JM, Maron DJ, Mackey SF, Superko HR, Williams PT, Johnstone IM, Champagne MA, Krauss RM, et al. Effects of intensive multiple risk factor reduction on coronary atherosclerosis and clinical cardiac events in men and women with coronary artery disease. The Stanford Coronary Risk Intervention Project (SCRIP). Circulation. 1994 Mar;89(3):975-90. doi: 10.1161/01.cir.89.3.975. PMID 8124838
- [Background] Quinn TG, Alderman EL, McMillan A, Haskell W. Development of new coronary atherosclerotic lesions during a 4-year multifactor risk reduction program: the Stanford Coronary Risk Intervention Project (SCRIP). J Am Coll Cardiol. 1994 Oct;24(4):900-8. doi: 10.1016/0735-1097(94)90848-6. PMID 7930223
- [Background] Miller BD, Alderman EL, Haskell WL, Fair JM, Krauss RM. Predominance of dense low-density lipoprotein particles predicts angiographic benefit of therapy in the Stanford Coronary Risk Intervention Project. Circulation. 1996 Nov 1;94(9):2146-53. doi: 10.1161/01.cir.94.9.2146. PMID 8901665